CLINICAL TRIAL: NCT05591131
Title: Genetic Testing in African Americans Towards Universal Paired Tumor/Germline Genetic Testing in Solid Tumor Patients With Specific Gynecological Malignancies
Brief Title: Genetic Testing in African Americans
Acronym: GTM-I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: GTM-I; Paceline (Other: GCC)
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Peritoneal Cancer
Keywords: Black and African American Health; Genetic Testing; Ovarian Cancer; Endometrial Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Time and Events Table (Experimental): Study Procedures are as followed:
  On Day 1 Surgery/biopsy will be performed to obtain ovarian and endometrial samples. Day 14 will include Informed consent, demographics collection and Blood samples will be obtained. Subjects will complete a survey about knowledge of, attitudes towards, and awareness of genetic testing use over 30 minutes on Day 14. Days 14-21 Tumor/blood DNA preparation. On Day 42 Genetic test results will be released and uploaded in the EMR. If the genetic testing is positive, genetic counseling will be scheduled.
  Interventions: Other: genetic testing; Other: Survey Administration

INTERVENTIONS:
Other: genetic testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Survey Administration — Complete survey

SUMMARY:
This is a pilot/feasibility study to conduct genetic testing using tumor/blood samples of African American and Caucasian patients with ovarian and endometrial cancer following surgery at AU Health Medical Center. The aim of the pilot/feasibility study is to sequence a panel of cancer genes on paired tumor/blood (germline) samples of patients with ovarian and endometrial tumors at a two-week time point following surgery at AU Medical Center. While paired testing of tumor and blood (germline) provides direct clinical value to patients, investigators propose to study whether investigators can define and overcome such minority barriers among the Georgia Cancer Center (GCC)/AU Health Medical Center (AUMC) patient population.

DETAILED DESCRIPTION:
The purpose of this study is to identify genetic mutations using a sequence a panel to detect cancer genes on paired tumor/blood (germline) samples particularly (AA) patients with ovarian, endometrial, fallopian or primary peritoneal carcinoma as AA individuals with cancer are less prone to accept a recommendation to undergo genetic testing. Approximately 30 subjects will participate in this study at Georgia Cancer Center/AU Health Medical Center.

Primary Objective:

To test the feasibility of this approach designed to provide a preliminary statistical analysis among the number of patients to overcome minority barriers among the GCC/AUMC patient population.

Secondary Objectives:

1. Measure attitudes toward early testing.
2. Compare rates of participation based on messaging of benefits between Caucasians and AA

Subjects must meet all inclusion criteria of the study. There are no exclusion criteria.

Patients will be identified by an AU Health gynecologic oncologist (SG, BR, RH). A research coordinator will be deployed to the clinic at the 2-week post-biopsy visit.

All subjects who consent to participate a clinical research coordinator will ask for their permission to provide a matched tumor and blood sample for genetic testing. If consented the subjects will be given a questionnaire regarding their knowledge of genetic testing for germline mutations. Tumor and blood samples will be collected for testing and sent to the Georgia Esoteric and Molecular Laboratory. It is estimated that it will take approximately one year to fully accrue and complete assessments on all participants entered on this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. New diagnosis of ovarian, endometrial, fallopian, or primary peritoneal carcinoma.
3. Diagnostic procedure performed at AU Health Medical Center.
4. Adequate tissue is available for the tumor testing component (e.g., cytology and FNA samples are typically not adequate, whereas core biopsies and open biopsies usually are adequate.
5. Consent at first post-biopsy outpatient clinic visit (typically about 2 weeks).
6. Ability to provide informed consent in English.

Exclusion Criteria:

There are no exclusion criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Consent rate for germline testing | 12 months
  Percentage of all patients with ovarian and endometrial cancer who complete testing

SECONDARY OUTCOMES:
Comparison of rate of Participation | 12 months
  Compare rates of participation based upon the patient's understanding the message regarding benefit and based upon her race.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Cancer Center at Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No